CLINICAL TRIAL: NCT00811109
Title: HEMOTOL: Effects of New Dialysis On-line Monitoring Devices on Hemodynamic Stability During Intermittent Hemodialysis in Critically Ill Patients With Acute Kidney Injury : a Prospective Randomized Study.
Brief Title: HEMOTOL: Efficacy and Safety of Hemodialysis On-line Monitoring Devices on Hemodynamic Stability in Intensive Care Unit
Acronym: HEMOTOL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: TERZI/MD, University Hospital, Caen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A08-D12-VOL.6
Record Dates: First submitted 2008-12-15; First posted 2008-12-18 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-03

CONDITIONS: Hemodialysis
Keywords: Acute Kidney Injury; Critical care; Hypotension; Renal replacement therapy; Efficacy; Tolerance; Outcome
MeSH Terms: conditions — Acute Kidney Injury; Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard (No Intervention): Gold standard bicarbonate hemodialysis therapy with constant ultrafiltration rate and dialysis conductivity
  Interventions: Device: Standard Hemodialysis
- 2 (Active Comparator): With Blood Volume on-line monitoring only
  Interventions: Device: with Blood Volume Management (BVM®) only
- 3 (Active Comparator): With Blood volume and Blood temperature on-line monitoring
  Interventions: Device: with Blood Volume (BVM®) and Temperature (BTM®) on-line monitoring

INTERVENTIONS:
Device: Standard Hemodialysis — Gold standard bicarbonate hemodialysis therapy with constant ultrafiltration rate and dialysis conductivity performed with Fresenius 4008S monitor (Fresenius Medical Care, France)
  Other Names: Treatment A
  Arms: Standard
Device: with Blood Volume Management (BVM®) only — Hemodialysis using Blood Volume on-line monitoring only. Hemodialysis will be performed with Fresenius 4008S monitor (Fresenius Medical Care, France) equipped with BVM® device (for blood volume monitor; Fresenius Medical Care, France)
  Other Names: Treatment B
  Arms: 2
Device: with Blood Volume (BVM®) and Temperature (BTM®) on-line monitoring — Hemodialysis using Blood volume and Blood temperature on-line monitoring. Hemodialysis will be performed with Fresenius 4008S monitor (Fresenius Medical Care, France) equipped with BVM® and BTM® devices (for blood volume monitor and blood temperature management, respectively; Fresenius Medical Care, France)
  Other Names: Treatment C
  Arms: 3

SUMMARY:
The purpose of this randomized controlled study is to compare the effects of different new dialysis on-line monitoring devices on hemodynamic stability during intermittent hemodialysis in critically ill patients with acute kidney injury.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is associated with high mortality and morbidity rates in critically ill patients despite advances in renal replacement therapy (RRT). Over the last few years, new devices in dialysis equipment, such as blood temperature and blood volume on-line monitors, have been developed to improve hemodynamic tolerance, and these new modalities have demonstrated their positive impact on decrease in intra-dialytic hypotension rate in chronic hemodialysis patients. In order to evaluate these new devices in critically ill patients with acute kidney injury we decided to conduct a prospective randomized controlled trial.

We based calculation of the sample size on a power analysis that assumed an expected decrease in intra-dialytic hypotension rate of 40% (from a crude intra-dialytic hypotension rate of 30% to 18%) in groups B and C, compared with group A. Analysis is done by intention to treat, according to prescribed new dialysis on-line monitoring devices.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute Kidney injury requiring intermittent hemodialysis

Exclusion Criteria:

* Age < 18 years
* End-stage renal failure
* Inclusion in other protocol
* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Intra-Dialytic Hypotension | 60 days

SECONDARY OUTCOMES:
Compliance to treatment; intra-dialytic complications; dialysis dose; blood temperature control; blood volume control | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Damien du CHEYRON, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Service de Réanimation Médicale - CHU de Caen, Caen, France

REFERENCES:
- [Derived] Marshall MR, Wang MY, Vandal AC, Dunlop JL. Low dialysate sodium levels for chronic haemodialysis. Cochrane Database Syst Rev. 2024 Nov 5;11(11):CD011204. doi: 10.1002/14651858.CD011204.pub3. PMID 39498822
- [Derived] du Cheyron D, Terzi N, Seguin A, Valette X, Prevost F, Ramakers M, Daubin C, Charbonneau P, Parienti JJ. Use of online blood volume and blood temperature monitoring during haemodialysis in critically ill patients with acute kidney injury: a single-centre randomized controlled trial. Nephrol Dial Transplant. 2013 Feb;28(2):430-7. doi: 10.1093/ndt/gfs124. Epub 2012 Apr 25. PMID 22535635